CLINICAL TRIAL: NCT00922402
Title: Heart & Diabetes - Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Heart & Diabetes
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-03

CONDITIONS: Acute Heart Failure
Keywords: Acute; heart failure; hyperglycemia; Acute heart failure with high levels of glycemia
MeSH Terms: conditions — Heart Failure; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): All patients will be submitted to a shared intensive protocol of insulin infusion supported by continuous glucose monitoring
  Interventions: Procedure: Intensive insulin infusion

INTERVENTIONS:
Procedure: Intensive insulin infusion — The intensive control of glycemia is obtained with a shared in-hospital insulin infusion protocol, supported by the use of a continuous glucose monitoring system (Medtronic Guardian REAL Time). Any sudden variation of glycemia levels and/or alarms, as indicated by the device, has to be confirmed with a finger-stick before any therapy modification.
  In-hospital management is subdivided in a 2-day intensive and a 3-day post-intensive phase.

SUMMARY:
The main purpose of this study is to validate an intensive protocol of insulin infusion and subsequent subcutaneous insulin administration with the support of continuous glucose monitoring, in addition to reference finger-stick values.

DETAILED DESCRIPTION:
Heart failure is a common disease (prevalence worldwide: 22 million; incidence worldwide: 2 million; prevalence in Italy: 750.000; incidence in Italy: 170.000), affecting 1-2% of overall population and accounting for a significant proportion of healthcare costs. Recurrent hospital admissions represent the majority of the disease-related cost. About 15-25% of patients with HF are diabetics: the presence of diabetes significantly worsens prognosis in patients with heart failure and increases the risk of death by 30% compared to subject without diabetes.

The intensive control of glycemia during acute heart failure is an objective of primary importance, which can be obtained only with a proper strategy of patient management and with a considerable organizational effort. In a shared protocol aimed at a tight control of glycemia, the use of Continuous Glucose Monitoring (CGM) is expected to allow an easier management of the patient and a more accurate implementation of the protocol.

The main purpose of this study is to validate an intensive protocol of insulin infusion and subsequent subcutaneous insulin administration with the support of continuous glucose monitoring, in addition to reference finger-stick values.

ELIGIBILITY:
Inclusion Criteria (all of the following inclusion criteria must be met for the patient to be enrolled in the study):

* acute heart failure, defined according to current ESC Guidelines
* HbA1c > 7.5% at admission in Cardiology Unit
* glycemia > 180 mg/dL at admission in Cardiology Unit
* the patients signed the Informed Consent

Exclusion Criteria (if any of the following criteria are met, patients cannot be enrolled in the study):

* heart failure in acute infarction or cardiogenic shock
* creatinemia > 3.5 mg/dL at admission or in hemodialytic therapy
* cirrhosis
* acute infective pathology
* cardiac revascularization during the hospitalization or in the preceding 3 months
* life expectance < 12 months
* age < 18 years
* pregnant women
* informed consent not signed
* subject included in other protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Average time to glycemic target (90-130 mg/dL) | Within two days after enrollment

SECONDARY OUTCOMES:
Number of patient-days without deviations from the protocol | Within two days after enrollment
Average glycemia in the first 6 hours | Within six hours after enrollment
Slope of decremental curve of glycemia in the first 6 hours | Within six hours after enrollment
Median number of glycemia controls/patient in the first 12 hours | Within twelve hours after enrollment
Percentage of patients in glycemic range during the first 6 hours of infusion | Within six hours after enrollment
Number of hypoglycemia episodes in the first 5 days | Within five days after enrollment
Number of medical interventions and/or therapy variations based on blood glucose monitoring (finger-sticks) and/or suggested by interstitial continuous glucose monitoring glucose monitoring in the first 5 days | Within five days after enrollment
HbA1c at 3 months and variation with respect to baseline | Within three months after enrollment
Number of hypoglycemia episodes in the follow-up | Within three months after enrollment
Evaluation of the number of finger-stick measurement and CGM readings | Within five days after enrollment
Evaluation of the correlation between finger-stick measurement and CGM readings | Within five days after enrollement
Number of times that therapy was changed after finger-stick confirmation when CGM values or alarms were indicating a therapy adjustment needs to be made | Within five days after enrollment
Number of times that finger-stick overruled CGM readings or alarms not to do any therapy adjustment | WIthin five days after enrollment
Evaluation of healthcare resource consumption | Within three months after enrollment
Evaluation of organizational impact | Within three months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Vigneri, MD, Study Chair — Garibaldi-Nesima Hospital - Catania - Italy; Maddalena Lettino, MD, Study Chair — Policlinico S. Matteo - Pavia - Italy; Michele Gulizia, MD, Study Chair — Garibaldi-Nesima Hospital - Catania - Italy; Luigi Magnani, MD, Study Chair — Policlinico S. Matteo - Pavia - Italy; Luigi Tavazzi, MD, Study Chair — Ospedale Villa Maria Cecilia - Gruppo Villa Maria - Cotignola (Ravenna) - Italy
Locations (2):
- Italy (2):
  - Garibaldi Nesima Hospital, Catania
  - Policlinico S. Matteo, Pavia